CLINICAL TRIAL: NCT04385329
Title: Shock Wave Therapy for Sural Myofascial Pain Syndrome Associated With Plantar Fasciitis: a Pilot Randomized Controlled Trial
Brief Title: Shock Wave Therapy for Sural Myofascial Pain Associated to Chronic Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Ettore Carlis, Physician specialised in physical medicine and rehabilitation, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160017179
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Tendinopathy
Keywords: Myofascial pain syndrome
MeSH Terms: conditions — Tendinopathy; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Experimental group:shock waves extended to gastrocnemius TrP (Experimental): Focused shock wave therapy was extended from the plantar fascia to the gastrocnemius-soleus trigger points.
  Interventions: Other: Shock wave therapy on plantar fascia extended to the gastrocnemius-soleus trigger points
- Control group: shock waves not extended to gastrocnemius TrP (Active Comparator): A standard focused shock wave therapy exclusively targeted at the plantar fascia
  Interventions: Other: Shock wave therapy on plantar fascia only

INTERVENTIONS:
Other: Shock wave therapy on plantar fascia extended to the gastrocnemius-soleus trigger points — Enrolled subjects were treated with focused shock wave therapy, once a week for three consecutive weeks, by a specialized physician with more than five years of expertise, using a device powered by a piezoelectric generator (PIEZOSON 100PLUS, Richard Wolf®). At each treatment session, with the patients lying in prone decubitus position, the enthesis of the plantar fascia and the gastrocnemius-soleus trigger points were clinically targeted and treated with a perpendicular technique.
  Arms: Experimental group:shock waves extended to gastrocnemius TrP
Other: Shock wave therapy on plantar fascia only — Enrolled subjects were treated with focused shock wave therapy, once a week for three consecutive weeks, by a specialized physician with more than five years of expertise, using a device powered by a piezoelectric generator (PIEZOSON 100PLUS, Richard Wolf®). At each treatment session, with the patients lying in prone decubitus position, the enthesis of the plantar fascia was clinically targeted and treated with a perpendicular technique.
  Arms: Control group: shock waves not extended to gastrocnemius TrP

SUMMARY:
The aim of this randomized controlled study in to investigate if a shock wave treatment extended to the gastrocnemius-soleus trigger points (TrP) is more effective than a standard treatment exclusively targeted at the plantar fascia in a population affected by unilateral plantar fasciitis with concomitant sural myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult age (18 to 75 years) and written informed consent;
* Unilateral heel pain of four weeks or longer duration;
* Pain to digital pressure in the insertional area of the plantar fascia at the calcaneum;
* Sonographic examination showing a plantar fascia thickness greater than 3.8mm (see procedures for details);
* Concomitant presence of a sural myofascial pain syndrome (SMPS), diagnosed on the basis of the finding, at the physical examination, of trigger points of the gastrocnemius-soleus muscle complex, according to Travel and Simons' original description.

Exclusion Criteria:

* No corticosteroid injections or other physical therapies since the onset of the current pain episode (except pharmacological pain treatments and foot orthoses);
* No general contraindication to shock wave therapy (pregnancy, bleeding disorders or anticoagulant drug usage, cancer in the focal area);
* No clinical signs of lumbar radiculopathy at physical examination;
* No ankle osteoarthritis, diagnosed on the basis of clinical and radiographic findings;
* No previous fractures or surgery in the affected ankle and foot;
* No rheumatologic diseases, no plantar fibromatosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Change in FFI-foot function index | FFI was administered at baseline, at two months time point and at three months time point
  Foot Function Index is self-administered questionnaire designed to measure foot performances in relation to symptoms. Foot Function Index is structured in two sections of nine items each, investigating foot pain (FFI-A) and function (FFI-B) respectively. The total score of each section ranges from zero (no pain/no functional limitation) to 100 (intolerable pain/complete inability). The two scores were separately analysed.

SECONDARY OUTCOMES:
Change in PPT-pressure pain threshold | PPT was recorded at baseline, at two months time point and at three months time point
  Pressure pain threshold (PPT) of the gastrocnemius-soleus trigger points was assessed by means of a digital hand-held algometer (see procedures for details). PPT is the minimal force that induces pain and its measurement is useful to quantitatively evaluate the effect of a treatment on trigger points

IPD SHARING:
Plan to Share IPD: No